CLINICAL TRIAL: NCT02276443
Title: ARTEMIS: A Robust TNBC Evaluation FraMework to Improve Survival
Brief Title: Molecular Testing and Imaging in Improving Response in Patients With Stage I-III Triple-Negative Breast Cancer Receiving Chemotherapy MDACC Breast Moonshot Initiative
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0185; NCI-2015-00191 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0185 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Invasive Breast Carcinoma; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Drug Therapy; Immunotherapy; Adjuvants, Immunologic; Sentinel Lymph Node Biopsy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (predictive results given) (Experimental): Patients undergo baseline molecular and IHC evaluation of their tumor biopsy, and receive the results. Patients then receive standard anthracycline-based chemotherapy and undergo standard ultrasound at baseline, after 2 cycles, after 4 cycles of treatment, and after completion of treatment (before surgery). Patients and physicians are notified of the results of the molecular evaluation. Patients may then choose to continue with standard taxane +/- platinum-based chemotherapy or participate in an experimental clinical trial designed to match the molecular profile and triple-negative subtype. Patients with tumors predicted to be insensitive to chemotherapy are advised to participate in a clinical trial treating their tumor subtype.
  Interventions: Drug: Chemotherapy; Other: Laboratory Biomarker Analysis; Procedure: Lymph Node Biopsy; Procedure: Ultrasonography
- Arm B (predictive results given) (Experimental): Patients undergo baseline molecular and IHC evaluation of their tumor biopsy, and receive the results. Patients then receive standard anthracycline-based chemotherapy and undergo standard ultrasound at baseline, after 2 cycles, and after 4 cycles of treatment. Patients and physicians are notified of the results of the molecular evaluation. Patients may then choose to continue with standard taxane +/- platinum-based chemotherapy or participate in an experimental clinical trial designed to match the molecular profile and triple-negative subtype. Patients with tumors predicted to be insensitive to chemotherapy are advised to participate in a clinical trial treating their tumor subtype.
  Interventions: Drug: Chemotherapy; Other: Laboratory Biomarker Analysis; Procedure: Lymph Node Biopsy; Procedure: Ultrasonography
- Arm C (predictive results given) (Experimental): Patients undergo baseline molecular and IHC evaluation of their tumor biopsy, and receive the results. Patients then receive standard anthracycline-based chemotherapy with immunotherapy and undergo standard ultrasound at baseline, after 2 cycles, and after 4 cycles of treatment. Patients and physicians are notified of the results of the molecular evaluation. Patients may then choose to continue with standard taxane +/- platinum-based chemotherapy or participate in an experimental clinical trial designed to match the molecular profile and triple-negative subtype. Patients with tumors predicted to be insensitive to chemotherapy are advised to participate in a clinical trial treating their tumor subtype
  Interventions: Drug: Chemotherapy; Other: Immunotherapy; Other: Laboratory Biomarker Analysis; Procedure: Lymph Node Biopsy; Procedure: Ultrasonography

INTERVENTIONS:
Drug: Chemotherapy — Receive standard chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Other: Immunotherapy — Receive standard immunotherapy
  Other Names: Immunological; Immunological Therapy; Immunologically Directed Therapy
  Arms: Arm C (predictive results given)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Lymph Node Biopsy — Undergo baseline lymph node evaluation
  Other Names: Biopsy of Lymph Node
Procedure: Ultrasonography — Undergo standard ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasound; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This clinical trial assesses whether a newly designed algorithm which looks at the genomic signature of each patient's tumor to predict their sensitivity to standard of care treatment verses being placed on a personally designed treatment trial can improve the responses in patients with newly diagnosed triple-negative breast cancer (TNBC). Testing the primary tumor biopsy for certain proteins and monitoring the lymphocyte infiltration into the tumors may help doctors determine the sub-type of TNBC, and direct treatments that may work well. It is not yet known whether assigning treatment based on the patient's tumor classification will improve how well the tumor responds.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To conduct a prospective single arm, non-randomized trial to determine the impact of implementation of a research platform that includes diagnostic imaging to assess response to the initial phase of neoadjuvant chemotherapy combined with subtyping of TNBC in order to select the appropriate targeted therapy trial to complete neoadjuvant chemotherapy in patients found to have chemo-insensitive disease by imaging.

SECONDARY OBJECTIVES:

I. Measured as defined by Standardized Definitions for Efficacy End Points (STEEP) criteria using the following prioritization: distant recurrence free interval (DRFI), recurrence free survival (RFS), distant relapse-free survival (DRFS), overall survival (OS), invasive disease free survival (IDFS), disease free survival including ductal carcinoma in situ (DFS-DCIS).

II. Evaluate the rates of enrollment into clinical trials for patients identified as having chemotherapy insensitive disease.

III. Evaluate the frequency of pathologic response rates (pCR, RCB I-III residual disease) in patients identified as chemotherapy sensitive versus insensitive.

IV. Determine the estimates of DRFI, RFS, DRFS, IDFS and DFS-DCIS at 3 years, and OS at 5 and 10 years in all patients.

X. Determine the pathologic response based on molecular characterization. XI. Determine the estimates of DRFI, RFS, DRFS, IDFS and DFS-DCIS at 3 years, and OS at 5 and 10 years.

XII. Subset analyses of pathologic response and 3-year DRFI, RFS, DRFS, IDFS, and DFS-DCIS.

XIII. Compare the results of pathologic node-negative status (sentinel and/or non-sentinel nodes) after neoadjuvant chemotherapy according to a genomic predictor of nodal response to NACT, in subsets defined by pre-treatment clinical nodal status.

EXPLORATORY OBJECTIVES:

I. Future re-analysis of residual samples using a customized genomic diagnostic platform (integrated "prospective-retrospective" biomarker analysis) to predict chemotherapy sensitivity.

II. Generation and subsequent molecular characterization of patient derived xenograph (PDX) models.

III. Clinical diagnostic development studies using residual samples (fresh and/or formalin-fixed) within the Clinical Laboratory Improvement Amendments (CLIA)-compliant Molecular Diagnostics Laboratory, and patient derived xenographs (PDX) to formally evaluate the clinical validity and utility of future clinical genomic diagnostic tests that would predict both response, recurrence, and survival from the treatments used in this clinical trial (correlative "retrospective-prospective" biomarker analyses).

IV. Correlative science studies to identify molecular therapeutic targets for treatment-insensitive TNBC using residual samples and PDX models.

V. Correlation of tumor features or changes as measured by diagnostic imaging to determine potential predictors of treatment response.

VI. Determine polymerase chain reaction (pCR) rates in a cohort of patients who undergo surgical resection after achieving complete radiological response after 4 cycles of adjuvant chemotherapy (AC).

OUTLINE: Patients are assigned to 1 of 3 arms.

ARM A: Patients undergo baseline molecular and immunohistochemistry (IHC) evaluation of their tumor biopsy, and receive the results. Patients then receive standard anthracycline-based chemotherapy and undergo standard ultrasound at baseline, after 2 cycles, after 4 cycles of treatment, and after completion of treatment (before surgery). Patients and physicians are notified of the results of the molecular evaluation. Patients may then choose to continue with standard taxane +/- platinum-based chemotherapy or participate in an experimental clinical trial designed to match the molecular profile and triple-negative subtype. Patients with tumors predicted to be insensitive to chemotherapy are advised to participate in a clinical trial treating their tumor subtype.

ARM B: Patients undergo baseline molecular and IHC evaluation of their tumor biopsy, and receive the results. Patients then receive standard anthracycline-based chemotherapy and undergo standard ultrasound at baseline, after 2 cycles, and after 4 cycles of treatment. Patients and physicians are notified of the results of the molecular evaluation. Patients may then choose to continue with standard taxane +/- platinum-based chemotherapy or participate in an experimental clinical trial designed to match the molecular profile and triple-negative subtype. Patients with tumors predicted to be insensitive to chemotherapy are advised to participate in a clinical trial treating their tumor subtype.

ARM C: Patients undergo baseline molecular and IHC evaluation of their tumor biopsy, and receive the results. Patients then receive standard anthracycline-based chemotherapy with immunotherapy and undergo standard ultrasound at baseline, after 2 cycles, and after 4 cycles of treatment. Patients and physicians are notified of the results of the molecular evaluation. Patients may then choose to continue with standard taxane +/- platinum-based chemotherapy or participate in an experimental clinical trial designed to match the molecular profile and triple-negative subtype. Patients with tumors predicted to be insensitive to chemotherapy are advised to participate in a clinical trial treating their tumor subtype.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient can undergo biopsy or surgery of a primary tumor site for suspected or proven invasive breast cancer of clinical stage I to III and are planned to receive neoadjuvant therapy with anthracycline/taxane based regimens (Arm A and Arm B) or chemotherapy/immunotherapy-based regimens (Arm C)
* The patient was proven to have TNBC, defined from standard pathologic assays as negative for ER and PR (< 10% tumor staining) and negative for HER2 (immunohistochemistry [IHC] score < 3, gene copy number not amplified)
* Patients must have left ventricular ejection fraction (LVEF) >= 50% by multi gated acquisition scan (MUGA) or echocardiogram (ECHO) within 12 weeks prior to starting adriamycin
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x institutional upper limit of normal
* Creatinine within 1.5 X the upper limits of normal OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* For Arms A and B, patients must be medically ineligible to receive immunotherapy in combination with anthracycline/taxane-based chemotherapy as part of standard care
* For Arm C, patients must be medically eligible to receive immunotherapy in combination with chemotherapy as part of standard of care

Exclusion Criteria:

* The patient has diagnosis of stage IV disease or is found to have stage IV disease prior to initiation of chemotherapy
* Prior history of invasive cancer within 5 years of study entry or history of metastatic cancer; exceptions include non-metastatic, curatively treated basal and squamous cell carcinoma of the skin
* Prior excisional biopsy of the primary invasive breast cancer
* Patients with hematomas or biopsy site changes that limit response assessment of the primary tumor by diagnostic imaging
* Patients not eligible for chemotherapy with taxane and/or anthracycline based chemotherapy regimens
* Prior therapy with - chemotherapy and/or immunotherapy
* Grade II or higher neuropathy
* Patients with Zubrod performance status of > 2
* Patients with history of serious cardiac events defined as:

  * Patients with a history of New York Heart Association class 3 or 4 heart failure, or history of myocardial infarction, unstable angina or cerebrovascular accident (CVA) within 6 months of protocol registration
  * Patients who have history of PR prolongation (grade 2 or higher) or atrioventricular (AV) block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 5 years
  A one-sided z-test will be used to compare the response rates of the treatment and control arms. The study will have 80% power to detect an increase in the response rate of 14.2 percentage points assuming a control arm response rate of 50% at the 0.05 significance level allowing for two interim tests for both futility and superiority.

SECONDARY OUTCOMES:
Survival | Up to 5 years
  Will estimate the cumulative incidence function using Aalen-Johansen method with appropriate 96% confidence intervals.
Frequency of tumors | Up to 5 years
  Will estimate the relative frequency to triple negative breast cancer (TNBC) subsets (BRCA+, mesenchymal, androgen receptor [AR]+ and basal-like) classified withing each predication cohort and report both point estimates and simultaneous multinomial 95% confidence intervals based on the method of Goodman.

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Yam, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- [Derived] Wang X, Zhao L, Song X, Wu X, Krishnamurthy S, Semba T, Shao S, Knafl M, Coffer LW 2nd, Alexander A, Vines A, Bopparaju S, Woodward WA, Chu R, Zhang J, Yam C, Loo LWM, Nasrazadani A, Huong LP, Woodman SE, Futreal A; Rare Tumor Initiative Team; Tripathy D, Ueno NT. Genomic and transcriptomic analyses identify distinctive features of triple-negative inflammatory breast cancer. NPJ Precis Oncol. 2024 Nov 18;8(1):265. doi: 10.1038/s41698-024-00729-0. PMID 39558017
- [Derived] Stowers CE, Wu C, Xu Z, Kumar S, Yam C, Son JB, Ma J, Tamir JI, Rauch GM, Yankeelov TE. Combining Biology-based and MRI Data-driven Modeling to Predict Response to Neoadjuvant Chemotherapy in Patients with Triple-Negative Breast Cancer. Radiol Artif Intell. 2025 Jan;7(1):e240124. doi: 10.1148/ryai.240124. PMID 39503605
- [Derived] Basho RK, Zhao L, White JB, Huo L, Bassett RL, Mittendorf EA, Thompson A, Litton JK, Ueno N, Arun B, Lim B, Valero V, Tripathy D, Zhang J, Adrada BE, Santiago L, Ravenberg E, Seth S, Yam C, Moulder SL, Damodaran S. Comprehensive Analysis Identifies Variability in PI3K Pathway Alterations in Triple-Negative Breast Cancer Subtypes. JCO Precis Oncol. 2024 Mar;8:e2300124. doi: 10.1200/PO.23.00124. PMID 38484209
- [Derived] Chen H, Ding Q, Khazai L, Zhao L, Damodaran S, Litton JK, Rauch GM, Yam C, Chang JT, Seth S, Lim B, Thompson AM, Mittendorf EA, Adrada B, Virani K, White JB, Ravenberg E, Song X, Candelaria R, Arun B, Ueno NT, Santiago L, Saleem S, Abouharb S, Murthy RK, Ibrahim N, Routbort MJ, Sahin A, Valero V, Symmans WF, Tripathy D, Wang WL, Moulder S, Huo L. PTEN in triple-negative breast carcinoma: protein expression and genomic alteration in pretreatment and posttreatment specimens. Ther Adv Med Oncol. 2023 Aug 2;15:17588359231189422. doi: 10.1177/17588359231189422. eCollection 2023. PMID 37547448
- [Derived] Hwang KP, Elshafeey NA, Kotrotsou A, Chen H, Son JB, Boge M, Mohamed RM, Abdelhafez AH, Adrada BE, Panthi B, Sun J, Musall BC, Zhang S, Candelaria RP, White JB, Ravenberg EE, Tripathy D, Yam C, Litton JK, Huo L, Thompson AM, Wei P, Yang WT, Pagel MD, Ma J, Rauch GM. A Radiomics Model Based on Synthetic MRI Acquisition for Predicting Neoadjuvant Systemic Treatment Response in Triple-Negative Breast Cancer. Radiol Imaging Cancer. 2023 Jul;5(4):e230009. doi: 10.1148/rycan.230009. PMID 37505106
- [Derived] Wu C, Jarrett AM, Zhou Z, Elshafeey N, Adrada BE, Candelaria RP, Mohamed RMM, Boge M, Huo L, White JB, Tripathy D, Valero V, Litton JK, Yam C, Son JB, Ma J, Rauch GM, Yankeelov TE. MRI-Based Digital Models Forecast Patient-Specific Treatment Responses to Neoadjuvant Chemotherapy in Triple-Negative Breast Cancer. Cancer Res. 2022 Sep 16;82(18):3394-3404. doi: 10.1158/0008-5472.CAN-22-1329. PMID 35914239
- [Derived] Yam C, Abuhadra N, Sun R, Adrada BE, Ding QQ, White JB, Ravenberg EE, Clayborn AR, Valero V, Tripathy D, Damodaran S, Arun BK, Litton JK, Ueno NT, Murthy RK, Lim B, Baez L, Li X, Buzdar AU, Hortobagyi GN, Thompson AM, Mittendorf EA, Rauch GM, Candelaria RP, Huo L, Moulder SL, Chang JT. Molecular Characterization and Prospective Evaluation of Pathologic Response and Outcomes with Neoadjuvant Therapy in Metaplastic Triple-Negative Breast Cancer. Clin Cancer Res. 2022 Jul 1;28(13):2878-2889. doi: 10.1158/1078-0432.CCR-21-3100. PMID 35507014
- [Derived] Yam C, Yen EY, Chang JT, Bassett RL, Alatrash G, Garber H, Huo L, Yang F, Philips AV, Ding QQ, Lim B, Ueno NT, Kannan K, Sun X, Sun B, Parra Cuentas ER, Symmans WF, White JB, Ravenberg E, Seth S, Guerriero JL, Rauch GM, Damodaran S, Litton JK, Wargo JA, Hortobagyi GN, Futreal A, Wistuba II, Sun R, Moulder SL, Mittendorf EA. Immune Phenotype and Response to Neoadjuvant Therapy in Triple-Negative Breast Cancer. Clin Cancer Res. 2021 Oct 1;27(19):5365-5375. doi: 10.1158/1078-0432.CCR-21-0144. PMID 34253579